CLINICAL TRIAL: NCT06959173
Title: Organoid-guided Personalized Treatment of Pleural Effusion
Status: Recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Qiming Wang, Professor, Henan Cancer Hospital
Other Study IDs: 2024-592
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer
Keywords: Lung Cancer (NSCLC), Pleural effusion, patient-derived organoids
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Pleural Effusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study is a single-arm, single-center clinical research that utilizes patient-derived tumor organoids to predict drug sensitivity, thereby assisting clinicians in formulating treatment plans to benefit lung cancer patients with pleural effusion.

This study is divided into three parts: acquisition of clinical samples from patients, in vitro organoid culture and drug sensitivity testing, and correlation of organoid sensitivity results with clinical medication guidance. Researchers obtained pre-treatment tissue samples and provided them to Suzhou Xianjue Biotechnology Co., Ltd. to establish organoid models. Once established, drug incubation was performed for sensitivity testing. Subsequently, treatment for malignant pleural effusion was guided based on drug sensitivity data.

DETAILED DESCRIPTION:
Research name：Organoid-guided personalized treatment of pleural effusion.

Intervention study: Not have.

Research design: The study is a single-arm, single-center clinical research that utilizes patient-derived tumor organoids to predict drug sensitivity, thereby assisting clinicians in formulating treatment plans to benefitlung cancer patients with pleural effusion.

This study is divided into three parts: acquisition of clinical samples from patients, in vitro organoid culture and drug sensitivity testing, and correlation of organoid sensitivity results with clinical medication guidance. Researchers obtained pre-treatment tissue samples and provided them to Suzhou Xianjue Biotechnology Co., Ltd. to establish organoid models. Once established, drug incubation was performed for sensitivity testing. Subsequently, treatment for malignant pleural effusion was guided based on drug sensitivity data.

Sample capacity: 20.

Purpose of research: The purpose of this study is to use the patient-derived organoid model for drug sensitivity testing, to explore the patient-derived organoids for drug sensitivity prediction, so as to achieve the benefit of lung cancer patients with pleural effusion.

Fundamental purpose: Assessment of the efficacy of pleural effusion therapy guided by patient-derived organoid drug sensitivity prediction.

Secondary purpose: Agreement of organoid drug prediction and actual clinical benefit.

Inclusion Criteria:

(1)18 years of age and above; (2) Understand and voluntarily sign the informed consent form (ICF), and have good compliance, and can cooperate with diagnosis and follow-up; (3)ECOG score 0-2; (4) Accompanied by malignant pleural effusion; Presence of at least one measurable lesion as assessed by the investigator;

Exclusion Criteria:

1. A history of malignant tumor in the past 5 years;
2. Complicated with serious complications, such as uncontrolled heart disease, severe arrhythmia requiring medical treatment, persistent watery diarrhea, etc.;
3. Pregnant or lactating female patients; Patients deemed unsuitable for participation in this study.

Study termination criteria: Reasons for subject withdrawal from the study may include:

1. The subject withdrew his informed consent. Subjects were free to terminate study participation at any time without being compromised in further treatment. If the subject withdraws informed consent, they will be asked in detail if they agree to participate in safety follow-up, continue efficacy assessment (if not progressing), and survival follow-up;
2. Subjects were lost to follow-up;
3. die;
4. Other reasons.

Visit the plan: Treatment follow-up for 2 years:

1. Follow-up visits are made every 8 weeks and ± 7 days within 1 year after enrollment (within 48 weeks);
2. Patients will be followed up every 12 weeks ± 7 days within the 1 to 2 years after enrollment (within weeks 49 to 96).

Statistical analysis: Data analysis will be performed using the SPSS statistical software.

ELIGIBILITY:
Inclusion Criteria:

(1)18 years of age and above; (2) Understand and voluntarily sign the informed consent form (ICF), and have good compliance, and can cooperate with diagnosis and follow-up; (3)ECOG score 0-2; (4) Accompanied by malignant pleural effusion; Presence of at least one measurable lesion as assessed by the investigator;

Exclusion Criteria:

1. A history of malignant tumor in the past 5 years;
2. Complicated with serious complications, such as uncontrolled heart disease, severe arrhythmia requiring medical treatment, persistent watery diarrhea, etc.;
3. Pregnant or lactating female patients; Patients deemed unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer with malignant pleural effusion
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 12 months
  Evaluation of therapeutic efficacy for pleural effusion: Objective Response Rate (ORR)

SECONDARY OUTCOMES:
Evaluation of efficacy in primary pulmonary lesions: Objective response rate (ORR) | up to 24 months
  Assessed by Investigator According to RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Porcel JM, Gasol A, Bielsa S, Civit C, Light RW, Salud A. Clinical features and survival of lung cancer patients with pleural effusions. Respirology. 2015 May;20(4):654-9. doi: 10.1111/resp.12496. Epub 2015 Feb 23. PMID 25706291
- [Background] Penz E, Watt KN, Hergott CA, Rahman NM, Psallidas I. Management of malignant pleural effusion: challenges and solutions. Cancer Manag Res. 2017 Jun 23;9:229-241. doi: 10.2147/CMAR.S95663. eCollection 2017. PMID 28694705
- [Background] Asciak R, Rahman NM. Malignant Pleural Effusion: From Diagnostics to Therapeutics. Clin Chest Med. 2018 Mar;39(1):181-193. doi: 10.1016/j.ccm.2017.11.004. Epub 2017 Dec 13. PMID 29433714
- [Background] Clive AO, Kahan BC, Hooper CE, Bhatnagar R, Morley AJ, Zahan-Evans N, Bintcliffe OJ, Boshuizen RC, Fysh ET, Tobin CL, Medford AR, Harvey JE, van den Heuvel MM, Lee YC, Maskell NA. Predicting survival in malignant pleural effusion: development and validation of the LENT prognostic score. Thorax. 2014 Dec;69(12):1098-104. doi: 10.1136/thoraxjnl-2014-205285. Epub 2014 Aug 6. PMID 25100651
- [Background] Terra RM, Dela Vega AJM. Treatment of malignant pleural effusion. J Vis Surg. 2018 May 22;4:110. doi: 10.21037/jovs.2018.05.02. eCollection 2018. PMID 29963399
- [Background] Hackner K, Errhalt P, Handzhiev S. Ratio of carcinoembryonic antigen in pleural fluid and serum for the diagnosis of malignant pleural effusion. Ther Adv Med Oncol. 2019 May 22;11:1758835919850341. doi: 10.1177/1758835919850341. eCollection 2019. PMID 31205509
- [Background] Gayen S. Malignant Pleural Effusion: Presentation, Diagnosis, and Management. Am J Med. 2022 Oct;135(10):1188-1192. doi: 10.1016/j.amjmed.2022.04.017. Epub 2022 May 14. PMID 35576996
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- [Background] Ferro A, Marinato GM, Mulargiu C, Marino M, Pasello G, Guarneri V, Bonanno L. The study of primary and acquired resistance to first-line osimertinib to improve the outcome of EGFR-mutated advanced Non-small cell lung cancer patients: the challenge is open for new therapeutic strategies. Crit Rev Oncol Hematol. 2024 Apr;196:104295. doi: 10.1016/j.critrevonc.2024.104295. Epub 2024 Feb 20. PMID 38382773
- [Background] He J, Huang Z, Han L, Gong Y, Xie C. Mechanisms and management of 3rd-generation EGFR-TKI resistance in advanced non-small cell lung cancer (Review). Int J Oncol. 2021 Nov;59(5):90. doi: 10.3892/ijo.2021.5270. Epub 2021 Sep 24. PMID 34558640
- [Background] Passaro A, Mok TSK, Attili I, Wu YL, Tsuboi M, de Marinis F, Peters S. Adjuvant Treatments for Surgically Resected Non-Small Cell Lung Cancer Harboring EGFR Mutations: A Review. JAMA Oncol. 2023 Aug 1;9(8):1124-1131. doi: 10.1001/jamaoncol.2023.0459. PMID 37166792
- [Background] Rosell R, Moran T, Queralt C, Porta R, Cardenal F, Camps C, Majem M, Lopez-Vivanco G, Isla D, Provencio M, Insa A, Massuti B, Gonzalez-Larriba JL, Paz-Ares L, Bover I, Garcia-Campelo R, Moreno MA, Catot S, Rolfo C, Reguart N, Palmero R, Sanchez JM, Bastus R, Mayo C, Bertran-Alamillo J, Molina MA, Sanchez JJ, Taron M; Spanish Lung Cancer Group. Screening for epidermal growth factor receptor mutations in lung cancer. N Engl J Med. 2009 Sep 3;361(10):958-67. doi: 10.1056/NEJMoa0904554. Epub 2009 Aug 19. PMID 19692684
- [Background] Castellanos E, Feld E, Horn L. Driven by Mutations: The Predictive Value of Mutation Subtype in EGFR-Mutated Non-Small Cell Lung Cancer. J Thorac Oncol. 2017 Apr;12(4):612-623. doi: 10.1016/j.jtho.2016.12.014. Epub 2016 Dec 23. PMID 28017789
- [Background] Shi Y, Au JS, Thongprasert S, Srinivasan S, Tsai CM, Khoa MT, Heeroma K, Itoh Y, Cornelio G, Yang PC. A prospective, molecular epidemiology study of EGFR mutations in Asian patients with advanced non-small-cell lung cancer of adenocarcinoma histology (PIONEER). J Thorac Oncol. 2014 Feb;9(2):154-62. doi: 10.1097/JTO.0000000000000033. PMID 24419411
- [Background] Zhuang X, Zhao C, Li J, Su C, Chen X, Ren S, Li X, Zhou C. Clinical features and therapeutic options in non-small cell lung cancer patients with concomitant mutations of EGFR, ALK, ROS1, KRAS or BRAF. Cancer Med. 2019 Jun;8(6):2858-2866. doi: 10.1002/cam4.2183. Epub 2019 Apr 24. PMID 31016879
- [Background] Skoulidis F, Heymach JV. Co-occurring genomic alterations in non-small-cell lung cancer biology and therapy. Nat Rev Cancer. 2019 Sep;19(9):495-509. doi: 10.1038/s41568-019-0179-8. Epub 2019 Aug 12. PMID 31406302
- [Background] Duma N, Santana-Davila R, Molina JR. Non-Small Cell Lung Cancer: Epidemiology, Screening, Diagnosis, and Treatment. Mayo Clin Proc. 2019 Aug;94(8):1623-1640. doi: 10.1016/j.mayocp.2019.01.013. PMID 31378236
- [Background] Travis WD, Brambilla E, Nicholson AG, Yatabe Y, Austin JHM, Beasley MB, Chirieac LR, Dacic S, Duhig E, Flieder DB, Geisinger K, Hirsch FR, Ishikawa Y, Kerr KM, Noguchi M, Pelosi G, Powell CA, Tsao MS, Wistuba I; WHO Panel. The 2015 World Health Organization Classification of Lung Tumors: Impact of Genetic, Clinical and Radiologic Advances Since the 2004 Classification. J Thorac Oncol. 2015 Sep;10(9):1243-1260. doi: 10.1097/JTO.0000000000000630. PMID 26291008
- [Background] Zheng RS, Chen R, Han BF, Wang SM, Li L, Sun KX, Zeng HM, Wei WW, He J. [Cancer incidence and mortality in China, 2022]. Zhonghua Zhong Liu Za Zhi. 2024 Mar 23;46(3):221-231. doi: 10.3760/cma.j.cn112152-20240119-00035. Chinese. PMID 38468501